CLINICAL TRIAL: NCT02827994
Title: Pain Neurophysiology Education and Exercise for Adolescents With Chronic Idiopathic Neck Pain: a School-based Pilot, Randomised and Controlled Study
Brief Title: Pain Neurophysiology Education and Exercise for Adolescents With Chronic Idiopathic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Dr, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCEDCSS_FMUP 5/2015
Record Dates: First submitted 2016-06-23; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education and exercise (Experimental): The intervention included neurophysiology of pain education and exercises.
  Interventions: Other: neurophysiology of pain education and exercises
- No intervention (No Intervention): This group received no intervention as participants were students that were not seeking treatment for their pain.

INTERVENTIONS:
Other: neurophysiology of pain education and exercises — Pain neurophysiology education covered the neurophysiology of pain, transition from acute to chronic pain and the nervous system ability to modulate the pain experience. It was delivered in small groups (4 to 7 participants). A total of 4 sessions were delivered over 4 weeks (1 session per week). Each session took between 45 minutes and 1 hour.
  Exercises were aimed at increasing the endurance and strength of the deep neck flexor and extensor muscles and of the scapular muscles delivered over 3 sessions (the first session covered pain neurophysiology education only). Each exercise was performed in 3 series of 10 repetitions. The number of exercises targeting the same group of muscles increased from one in the 2nd session to 2/3 in the 4th session.
  Arms: Education and exercise

SUMMARY:
This study compared the effectiveness of pain neurophysiology education and neck/shoulder exercises with no intervention in adolescents with chronic idiopathic neck pain (CINP).

DETAILED DESCRIPTION:
Forty three adolescents with chronic idiopathic neck pain were randomly allocated to receive pain neurophysiology education and shoulder/neck exercises (n=21) or no intervention (n=22). Data on pain intensity (Visual Analogue Scale), pain disability, neck flexor and extensor muscles endurance, scapulae stabilizers endurance, pain catastrophizing (Pain catastrophizing Scale), trait and state anxiety (State-Trait Anxiety Inventory) and knowledge of pain neurophysiology (Neurophysiology of Pain Questionnaire) were collected. Measurements were taken before and after the intervention.

Statistical analysis were performed using a mixed-methods ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* To be invited to enter the study participants had to have chronic idiopathic neck/shoulder pain, defined as pain felt in the neck/shoulder regions at least once a week in the previous 3 months.

Exclusion Criteria:

* No exclusion criteria

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity | At the beginning
  Method of assessment - Visual analogue scale
Pain intensity | 5 weeks
  Method of assessment - Visual analogue scale

SECONDARY OUTCOMES:
Neck pain frequency | At the beginning
  Method of assessment - a question on neck pain frequency in the previous week (never, seldom, occasionally, often, always)
Neck pain frequency | 5 weeks
  Method of assessment - a question on neck pain frequency in the previous week (never, seldom, occasionally, often, always)
Neck pain duration | At the beginning
  Method of assessment - a question on neck pain duration (how long have you have neck pain?)
Neck pain duration | 5 weeks
  Method of assessment - a question on neck pain duration (how long have you have neck pain?)
Neck pain associated disability | At the beginning
  Method of assessment - a disability index with 5 questions on neck pain associated disability
Neck pain associated disability | 5 weeks
  Method of assessment - a disability index with 5 questions on neck pain associated disability
Neck flexor muscles endurance test | At the beginning
  Method of assessment - physical test; the participant is in supine and he/she is asked to flex the upper cervical spine, move their head away from the couch approximately 2.5 cm and then maintain this position for as long as possible. The test result is the time (in seconds) that each participant holds the position.
Neck flexor muscles endurance test | 5 weeks
  Method of assessment - physical test; the participant is in supine and he/she is asked to flex the upper cervical spine, move their head away from the couch approximately 2.5 cm and then maintain this position for as long as possible. The test result is the time (in seconds) that each participant holds the position.
Neck extensor muscles endurance test | At the beginning
  Method of assessment - physical test; the participant is in prone and position, head neutral, and supporting 2 Kg weight hanging from it. Participants were asked to support this weight for as long as possible while maintaining the neutral head positioning. The test result is the time (in seconds) that each participant holds the position.
Neck extensor muscles endurance test | 5 weeks
  Method of assessment - physical test; the participant is in prone and position, head neutral, and supporting 2 Kg weight hanging from it. Participants were asked to support this weight for as long as possible while maintaining the neutral head positioning. The test result is the time (in seconds) that each participant holds the position.
Scapular stabilizers' endurance test | At the beginning
  Method of assessment - physical test; Method of assessment - physical test; Participants were standing with the shoulders and elbows flexed at 90º, while pulling both extremities of a dynamometer to reach 1 Kg of force. The test result is the time (in seconds) that each participants was able to hold this position.
Scapular stabilizers' endurance test | 5 weeks
  Method of assessment - physical test; Method of assessment - physical test; Participants were standing with the shoulders and elbows flexed at 90º, while pulling both extremities of a dynamometer to reach 1 Kg of force. The test result is the time (in seconds) that each participants was able to hold this position.
State-trait anxiety inventory | At the beginning
  Method of assessment - scale
State-trait anxiety inventory | 5 weeks
  Method of assessment - scale
Pain Catastrophizing Scale | At the beginning
  Method of assessment - scale
Pain Catastrophizing Scale | 5 weeks
  Method of assessment - scale
Neurophysiology of pain questionnaire | At the beginning
  Method of assessment - questionnaire
Neurophysiology of pain questionnaire | 5 weeks
  Method of assessment - questionnaire
Patients' Global Impression of Change | 5 weeks
  Method of assessment - scale

IPD SHARING:
Plan to Share IPD: No